CLINICAL TRIAL: NCT03557983
Title: Evaluation of Fenofibrate on Radiation-induced Skin Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, zhangshuyu, Shuyu Zhang Associate Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SoochowU
Record Dates: First submitted 2018-05-19; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Radiodermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Fenofibrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fenofibrate (Experimental): Fenofibrate should be topically spread three times per day at the irradiated areas, with a concentration of 400 μg/mL for week.
  Interventions: Drug: Fenofibrate
- Saline (Placebo Comparator): Saline is topically spread three times per day for one week.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate is dissolved in Saline and topically spread three times per day at the irradiated areas, with a concentration of 400 μg/mL for week.
  Arms: fenofibrate
Drug: Saline — Saline is topically spread three times per day at the irradiated areas for one week.
  Arms: Saline

SUMMARY:
Fenofibrate is a specific ligand for PPARα, which has been used for the treatment of hypercholesterolemia, hypertriglyceridemia, diabetes and cardiovascular diseases for long time. Fenofibrate reduces low-density lipoprotein (LDL), very low density lipoprotein (VLDL) and triglyceride levels, while increases high-density lipoprotein (HDL) levels. PPARα has also shown antioxidant and anti-inflammatory properties. Fenofibrate confers cytoprotective effect against myocardial ischemia-reperfusion (I/R) injury in rats by suppressing cell apoptosis and ameliorates age-related renal injury through the activation of AMPK and SIRT1 signaling. However, the safety and effectiveness of fenofibrate on the progression of radiation-induced skin injury remain unknown. The purpose of this study is to determine whether topical application of fenofibrate is safe and effective for radiation-induced skin injury.

DETAILED DESCRIPTION:
Radiation-induced skin injury is a significant side effect of ionizing radiation delivered to the skin during cancer treatment as well as a result of other exposure to radiation. The skin is one of radiosensitive organ systems in human body because it is a continuously renewing organ containing rapidly proliferating and maturing cells. Ionizing radiation promotes reactive nitrogen and oxygen species (RNS/ROS) production due to radiolysis of water and direct ionization of target molecules, which result in oxidative damage and skin injuries. It is considered that ~95 % of cancer patients receiving radiation therapy will develop some form of radiodermatitis, including erythema, dry desquamation, and moist desquamation. Radiation-induced skin injury negatively affects the process of radiotherapy and the quality of patients' life. Despite substantial improvements in radiation technology, radiation-induced skin toxicity is still a concerning problem. The purpose of this study is to determine whether topical application of fenofibrate is safe and effective for radiation-induced skin injury.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients had to have a pathologically proven cancer with a planned course of radiotherapy.
* Normal haematological function (granulocyte count > 1.5 X 109 cells per litre, platelet count > 100 X 109 cells per litre and haemoglobin > 100 g/L) and organ function (creatinine clearance > 50 mL/min) and aspartate aminotransferase/alanine aminotransferase < 2.5 of upper normal limit).

Exclusion Criteria:

* The presence of rash or unhealed wound in the radiation field, known allergy or hypersensitivity to fenofibrate, pregnancy or lactation, history of/current connective tissue disorder and prior radiation to the thorax.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-13 (Estimated); Primary Completion 2020-04-13 (Estimated); Study Completion 2020-04-13 (Estimated)

PRIMARY OUTCOMES:
Measurement of skin wound area | 3 months
  Skin wound area was measured by software-based analysis.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Fenofibrate | 3 months
  Toxicity of Fenofibrate was graded using the NCI Common Terminology Criteria for Adverse Events v. 3.0. Any adverse event. Grade 1 attributed to fenofibrate was considered dose-limiting toxicity (DLT).
Evaluation of skin injury | 2 week
  Skin toxicity of radiotherapy was evaluated every day, once radiation began. Fenofibrate administration was given immediately when Grade 1 dermatitis occurred, and then dermatitis was recorded weekly. The score at the end of radiotherapy was the one of the last week of radiotherapy. The evaluation continued until 2 weeks after the end of radiotherapy with two approaches. The standard was the RTOG score defined by the observers.
Evaluation of skin toxicity of radiotherapy | 2 week
  Skin toxicity of radiotherapy was evaluated every day, once radiation began. Fenofibrate administration was given immediately when Grade 1 dermatitis occurred, and then dermatitis was recorded weekly. The score at the end of radiotherapy was the one of the last week of radiotherapy. The evaluation continued until 2 weeks after the end of radiotherapy with two approaches. Patient-reported symptom scores was adapted from the Skin Toxicity Assessment Tool as pain, burning, itching, pulling and tenderness in the treatment area.

CONTACTS AND LOCATIONS:
Overall Officials: Shuyu Zhang, A/Prof., Principal Investigator — Soochow University
Locations (1):
- 苏州大学, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao Q, Cui Z, Zheng Y, Li Q, Xu C, Sheng X, Tao M, Xu H. Fenofibrate protects against acute myocardial I/R injury in rat by suppressing mitochondrial apoptosis as decreasing cleaved caspase-9 activation. Cancer Biomark. 2017 Jul 4;19(4):455-463. doi: 10.3233/CBM-170572. PMID 28582851
- [Background] Kim EN, Lim JH, Kim MY, Kim HW, Park CW, Chang YS, Choi BS. PPARalpha agonist, fenofibrate, ameliorates age-related renal injury. Exp Gerontol. 2016 Aug;81:42-50. doi: 10.1016/j.exger.2016.04.021. Epub 2016 Apr 27. PMID 27130813
- [Background] Liu J, Lu C, Li F, Wang H, He L, Hao Y, Chen AF, An H, Wang X, Hong T, Wang G. PPAR-alpha Agonist Fenofibrate Upregulates Tetrahydrobiopterin Level through Increasing the Expression of Guanosine 5'-Triphosphate Cyclohydrolase-I in Human Umbilical Vein Endothelial Cells. PPAR Res. 2011;2011:523520. doi: 10.1155/2011/523520. Epub 2011 Nov 16. PMID 22190909